CLINICAL TRIAL: NCT03933189
Title: Physical Therapy for Individuals With Chronic Pain Due to Physical and/or Emotional Trauma: A Comparison of Physical Therapy Interventions
Brief Title: Physical Therapy to Treat Chronic Pain in Survivors of Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Justine Dee, Clinical Associate Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00000128
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain; Disability Physical
Keywords: chronic pain; trauma; rehabilitiation; physical therapy; musculoskeletal pain
MeSH Terms: conditions — Chronic Pain; Wounds and Injuries; Musculoskeletal Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Blinded randomized controlled study.
Who Masked: Outcomes Assessor
Masking Description: Participants will complete all the research outcome measures with a blinded independent examiner who will not be treating the participants and who will not know which treatment group participants are randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomedical (BIOM) physical therapy (Active Comparator): Six 60 minute PT sessions consisting of 15 minutes of education on topics such as ideal postural alignment (sitting, sleeping), maintenance of normal spinal curves, body mechanics, proper lifting techniques, home pain control via anti-inflammatory modalities such as ice; 15 minutes of manual therapy to region of pain (soft tissue and/or joint mobilization); 30 minutes of region specific exercises to address identified muscle imbalances -stretching and strengthening of the muscles local to the area of pain.
  Interventions: Other: Physical Therapy
- Biopsychosocial (BPS) physical therapy (Active Comparator): Six 60 minute PT sessions consisting of 15 minutes of pain neuro-science education, 15 minutes of Graded Motor Imagery (GMI) techniques, (a progressive program of visual and mental exercises consisting of laterality exercises, motor imagery and mirror therapy); 30 minutes of a general conditioning exercise program individualized for each participant based on initial examination findings and participant presentation consisting of:
  A cardiovascular component which may include walking on a treadmill, stationary cycling, or a seated stepping machine.
  A muscle strengthening component for extremities and trunk. A flexibility component for upper and lower extremity musculature.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical therapy modalities to treat chronic pain

SUMMARY:
This study will assess the effects of physical therapy (PT) for individuals who are survivors of trauma (SOT) and have chronic pain. While much has been studied about the psychological effects and treatment of trauma, little is known about the PT management of chronic pain and loss of function SOT experience. With over 24 million people in the U.S. suffering from chronic pain there are potentially high numbers of individuals living with resultant disability associated with that pain. Physical therapists are well versed in treating pain and restoring function. However, choice of PT can vary based on therapist years of experience and type or lack of PT specialization. Physical therapy has traditionally focused on a bio-medical (BIOM) approach. Some believe that the BIOM approach is ineffective in reducing chronic pain and functional loss, and that PT requires a biopsychosocial (BPS) approach, targeting central nervous system changes that occur with chronic pain. Pain education (PE) and Graded Motor Imagery (GMI) are PT interventions thought to address these brain changes, and are used by physical therapists to treat patients with phantom limb pain and Complex Regional Pain Syndrome. Most of the studies examining the effects of GMI and PE have methodological issues. Exercise is another common PT treatment and is beneficial in promoting improved function and decreasing disability for many conditions. Although PTs in clinical practice can offer all of these modalities, there is little high quality evidence to support the choice among them. This study will compare two varieties of PT: BIOM-based versus BPS-based care. Individuals with chronic pain who are referred to PT by their primary care provider or self-referred will be screened for trauma history by the PI. SOT who are seen at a community psychology center who experience chronic pain and disability will be referred to PT. Upon referral, SOT who meet the inclusion criteria will be invited to participate. SOT who consent to the study will be randomized to either the BIOM-based or the BPS-based group. All participants will undergo baseline assessment. Participants will complete 6 one-hour PT sessions once a week following their randomly assigned plan. All baseline measures will be repeated by the blinded assessor after the 6th visit; scores will be assessed to determine if there is a difference in the change in functional outcomes between the BIOM- and BPS-based groups after completion of the 6 PT sessions.

DETAILED DESCRIPTION:
The purpose of this study is to compare two usual PT programs to determine if one is more effective than the other in reducing disability and pain in individuals who are survivors of physical and or emotional trauma. Numerous studies have assessed the mental health issues of SOT and the psychological interventions used to address these issues, but there has been little research on interventions that address the somatic pain and disability complaints in SOT in spite of the fact that 78-83% of survivors report chronic pain.

There is large variability in physical therapy management of painful conditions, representing an opportunity to improve patient care and outcomes. Choice of physical therapy intervention can vary based on the individual therapist's years of experience or type of PT practice specialization, or lack of specialization. The biomedical model (BIOM) of physical therapy (PT) management addresses pain problems by targeting treatment towards the physiologic structures or tissues in the region where the patient is reporting the pain sensations. This model follows the premise that pain is due to tissue damage and localized inflammation due to faulty biomechanics and movement patterns, injury, disease or disuse. The Academy of Orthopedic Physical Therapists Low Back Pain Clinical Practice Guidelines recommend manual therapy, targeted spine strengthening, endurance and flexibility exercises to treat patients with acute, sub-acute, and chronic back pain, and follows this BIOM approach. Additionally, there are a variety of exercise methods and manual therapies touted by practitioners leading to heterogeneous interventions given for similar patient conditions. A 2014 study compared the outcomes of two different types of targeted spine interventions for the treatment of low back pain, and found the results to be equivocal, with approximately half the subjects in each treatment group demonstrating significant improvement. A biopsychosocial (BPS) PT approach of pain neuroscience education, Graded Motor Imagery and general conditioning exercises encompassing the health and skill related components of fitness has also been found to reduce pain and improve function in patients with chronic low back pain, in patients with complex regional pain syndrome and in patients with phantom limb pain. These conditions involve central brain changes due to the experience of chronic pain; pain neuroscience education and Graded Motor Imagery are purported to address these central changes. These studies, however, had methodologic issues, such as lack of a control group or small sample sizes. Exercise helps address the fear avoidance component of chronic low back pain, and helps to improve strength, endurance and tolerance for daily functional activities. Furthermore, pain education was found to decrease pain and improve function in SOT in a small pilot study. Patient education is a major component of any PT intervention.

There are a few small studies that have examined the effects of a BPS approach with promising results for specific chronic pain conditions, and there are studies that support the BIOM approach in treating musculoskeletal pain conditions but BPS- and BIOM-based treatments have not previously been compared in a large randomized controlled trial, nor described in the treatment of chronic pain in STT.

Researchers have sought to determine PT methods that are most beneficial in reducing chronic pain and disability, but studies to date have been inconclusive. The investigators objective is to compare the BIOM and BSP methods of PT to identify best treatment for individuals who have experienced physical and/or emotional trauma and have resultant disabling chronic pain due to this trauma. Findings from this work could help physical therapists provide targeted, effective treatment to help ameliorate the effects of chronic pain and disability in this population. With 78-83% of SOT living with chronic pain, the study findings will help therapists choose appropriate interventions to achieve optimal patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* definition of trauma/torture as defined by the United Nations (UN) HUR 03051 determined by referring clinical psychologist
* definition of trauma as identified through screening via the Life Events Check List by the PI
* chronic spine and or extremity pain of greater than 6 months duration
* able to attend and participate in six, 60-minute intervention sessions
* ambulatory, with or without assistive devices for a minimum of 20 feet

Exclusion Criteria:

* Inability to walk a minimum of 20 feet
* inability to afford any insurance fee for the 6 visits needed for the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) Computer Adaptive Test (CAT) | Baseline (pre-PT, week 0) and after completion of the 6th PT visit, at week 6
  Self report tool assessing physical function using a 5 point scale ranging from "1 Unable to do" to "5 Without any difficulty". Values are summed into a raw score, which is converted into a T-score. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference (PI) Computer Adaptive Test (CAT) | Baseline (pre-PT, week 0) and after completion of the 6th PT visit, at week 6
  Self report tool assessing how pain interferes and hinders engagement with social, cognitive, emotional, physical and recreational activities using a 5 point scale ranging from "1 Not at All", "2 A little bit", "3 Some what", "4 Quite a bit", "5 very much". Values are summed into a raw score, which is converted into a T-score. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) 29 | Baseline (pre-PT, week 0) and after completion of the 6th PT visit, at week 6.
  Self report tool assessing physical, mental, social health and wellbeing domains. Domains are scored on a 1-5 scale. Physical function scale ranges from "1 Unable to do" to "5 Without any difficulty"; anxiety, depression and ability to participate in social roles domain scales ranges from "1 Never" to "5 Always"; Fatigue, Sleep and Pain Interference domain scales range from "1 Not at all" to "5 Very Much" Values are summed into a raw score, which is converted into a T-score The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Change in Brief Pain Inventory | Baseline (pre-PT, week 0) and after completion of the 6th PT visit, at week 6
  Self report tool assessing pain intensity on an 11 point scale ranging from "0 No Pain" to "10 Pain as bad as you can imagine" and pain interference on an 11 point scale ranging from "0 Does not interfere" to "10 Completely Interferes". The 4 Pain intensity scores are used singly to represent pain severity. The Pain Interference is scored as the mean of the 7 items.
Change in Central Sensitization Inventory | Baseline (pre-PT, week 0) and after completion of the 6th PT visit, at week 6.
  Self report screening tool to identify central sensitization syndromes, measuring a participants self reported sensitivity to stimuli such as light, sounds, smells, muscle input and activity, on a 5 point scale ranging from "0 Never" to "4 Always". Values are summed into a total score, with higher score being worse sensitivity.
Change in Pain pressure threshold sensory testing | Baseline (pre-PT, week 0) and after completion of the 6th PT visit, at week 6.
  Quantitative sensory assessment of an individuals threshold to an applied pressure
Change in Two-point discrimination sensory testing | Baseline (pre-PT, week 0) and after completion of the 6th PT visit, at week 6.
  Quantitative sensory assessment of an individuals ability to discern one or two points of sensory input

CONTACTS AND LOCATIONS:
Overall Officials: Justine Dee, MS, Principal Investigator — University of Vermont
Locations (1):
- Dee Physical Therapy, South Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Williams AC, Pena CR, Rice AS. Persistent pain in survivors of torture: a cohort study. J Pain Symptom Manage. 2010 Nov;40(5):715-22. doi: 10.1016/j.jpainsymman.2010.02.018. Epub 2010 Aug 3. PMID 20678891
- [Result] Baird E, Williams ACC, Hearn L, Amris K. Interventions for treating persistent pain in survivors of torture. Cochrane Database Syst Rev. 2017 Aug 18;8(8):CD012051. doi: 10.1002/14651858.CD012051.pub2. PMID 28820231
- [Result] Kim HJ, Yu SH. Effects of complex manual therapy on PTSD, pain, function, and balance of male torture survivors with chronic low back pain. J Phys Ther Sci. 2015 Sep;27(9):2763-6. doi: 10.1589/jpts.27.2763. Epub 2015 Sep 30. PMID 26504288
- [Result] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Result] Henry SM, Van Dillen LR, Ouellette-Morton RH, Hitt JR, Lomond KV, DeSarno MJ, Bunn JY. Outcomes are not different for patient-matched versus nonmatched treatment in subjects with chronic recurrent low back pain: a randomized clinical trial. Spine J. 2014 Dec 1;14(12):2799-810. doi: 10.1016/j.spinee.2014.03.024. Epub 2014 Mar 22. PMID 24662210
- [Result] Moseley GL, Flor H. Targeting cortical representations in the treatment of chronic pain: a review. Neurorehabil Neural Repair. 2012 Jul-Aug;26(6):646-52. doi: 10.1177/1545968311433209. Epub 2012 Feb 13. PMID 22331213
- [Result] Malfliet A, Kregel J, Meeus M, Danneels L, Cagnie B, Roussel N, Nijs J. Patients With Chronic Spinal Pain Benefit From Pain Neuroscience Education Regardless the Self-Reported Signs of Central Sensitization: Secondary Analysis of a Randomized Controlled Multicenter Trial. PM R. 2018 Dec;10(12):1330-1343.e1. doi: 10.1016/j.pmrj.2018.04.010. Epub 2018 May 9. PMID 29753112
- [Result] Simons LE, Elman I, Borsook D. Psychological processing in chronic pain: a neural systems approach. Neurosci Biobehav Rev. 2014 Feb;39:61-78. doi: 10.1016/j.neubiorev.2013.12.006. Epub 2013 Dec 27. PMID 24374383
- [Result] Bowering KJ, O'Connell NE, Tabor A, Catley MJ, Leake HB, Moseley GL, Stanton TR. The effects of graded motor imagery and its components on chronic pain: a systematic review and meta-analysis. J Pain. 2013 Jan;14(1):3-13. doi: 10.1016/j.jpain.2012.09.007. Epub 2012 Nov 15. PMID 23158879
- [Result] Daffada PJ, Walsh N, McCabe CS, Palmer S. The impact of cortical remapping interventions on pain and disability in chronic low back pain: a systematic review. Physiotherapy. 2015 Mar;101(1):25-33. doi: 10.1016/j.physio.2014.07.002. Epub 2014 Aug 1. PMID 25442672
- [Result] Flor H, Denke C, Schaefer M, Grusser S. Effect of sensory discrimination training on cortical reorganisation and phantom limb pain. Lancet. 2001 Jun 2;357(9270):1763-4. doi: 10.1016/S0140-6736(00)04890-X. PMID 11403816
- [Result] Wallman KE, Morton AR, Goodman C, Grove R, Guilfoyle AM. Randomised controlled trial of graded exercise in chronic fatigue syndrome. Med J Aust. 2004 May 3;180(9):444-8. doi: 10.5694/j.1326-5377.2004.tb06019.x. PMID 15115421
- [Result] Landmark T, Romundstad P, Borchgrevink PC, Kaasa S, Dale O. Associations between recreational exercise and chronic pain in the general population: evidence from the HUNT 3 study. Pain. 2011 Oct;152(10):2241-2247. doi: 10.1016/j.pain.2011.04.029. Epub 2011 May 23. PMID 21601986